CLINICAL TRIAL: NCT05879432
Title: Phase 2 Global, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of LSALT Peptide for the Prevention or Attenuation of Acute Kidney Injury (AKI) in Patients Undergoing On-Pump Cardiac Surgery
Brief Title: LSALT Peptide for Prevention or Attenuation of Acute Kidney Injury (AKI) in Patients Undergoing On-Pump Cardiac Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arch Biopartners Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: AB003
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LSALT Peptide (Experimental): LSALT peptide 10 mg IV administered over 1 hour twice daily, every 12 ± 1 hour, for 5 days
  Interventions: Drug: LSALT Peptide
- Placebo (Placebo Comparator): Placebo IV administered over 1 hour twice daily, every 12 ± 1 hour, for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LSALT Peptide — LSALT, a peptide drug with the sequence NH3-LSALTPSPSWLKYKAL-COOH, binds to dipeptidase-1 (DPEP-1) but does not inhibit its biologic enzymatic activity, potentially minimizing off-target or other adverse effects. LSALT peptide inhibits leukocyte recruitment in multiple experimental disease models through the direct inhibition of leukocyte adhesion to DPEP-1 present in lungs, kidney, and liver.
  Other Names: Metablok
  Arms: LSALT Peptide
Drug: Placebo — 0.9% saline solution
  Arms: Placebo

SUMMARY:
To evaluate the percentage of subjects with AKI within 7 days following on-pump cardiac surgery defined by the KDIGO (Kidney Disease: Improving Global Outcomes) criteria:

1. Increase in baseline (pre-surgery) serum creatinine (SCr) by ≥26.5 μmol/L (≥0.3 mg/dL) within 7 days; OR
2. Increase in baseline SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the first 7 days following surgery; OR
3. Urine output < 0.5 mL/kg/h for >6 hours.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multicenter interventional study to assess safety and efficacy of LSALT peptide versus placebo (matching drug-free saline) in patients undergoing on-pump cardiac surgery. Patients will be followed for safety and efficacy up to Day 28 (EOS), with Day 1 being the day of randomization of study drug administered at least 1 hour prior to induction of anesthesia.

A total of 240 patients will be included in the study, 120 patients each will be randomized to LSALT peptide or placebo. This study will be double-blinded with only the pharmacist at the site unblinded for the purpose of preparing drug/placebo for injection.

All subjects will undergo tests during the Screening period (window days -14 to Day 1). After satisfying all inclusion and exclusion criteria, the patient will be randomized equally to the following study arms:

* LSALT peptide 10 mg IV administered over 1 hour twice daily, every 12 ± 1hour, for 5 days
* Placebo IV administered over 1 hour twice daily, every 12 ± 1 hour, for 5 days

Study treatment will be initiated pre-operatively on Day 1 and continued for 5 days. Physical examinations, vital signs and urine output will be recorded daily throughout the treatment period and on days 6 and 7. Adverse events will be recorded daily throughout the treatment period, on Days 6, 7, and 28 EOS (Day 28). Kidney function (serum creatinine, serum cystatin C, and BUN), clinical laboratory tests, and other biomarkers will be assessed at baseline (prior to initiation of study drug) and monitored daily throughout the treatment period, on Days 6, 7, and EOS (Day 28). All patients will be maintained on the standard of care (SOC) as per institutional guidelines. Thus, SOC will be followed in each patient with the addition of LSALT peptide or placebo.

Subjects will be followed until EOS (Day 28 ± 3 days) to assess renal function as discussed above.

An independent Data and Safety Monitoring Board (DSMB) will evaluate patients on a continuing basis for primarily safety assessments. Per the DSMB Charter, the DSMB will meet at least monthly if not more frequently based upon enrollment throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years of age.
2. Scheduled for a non-emergent coronary and/or valve surgery procedure requiring on-pump cardiopulmonary bypass including but not limited to:

   * Coronary artery bypass graft (CABG) alone
   * CABG with aortic, mitral, tricuspid, or pulmonic valve replacement or repair
   * Aortic valve replacement or repair alone, with or without aortic root repair
   * Mitral, tricuspid, or pulmonic valve replacement or repair alone
   * Simultaneous replacement of several cardiac valves.
3. Have the following AKI risk factors:

   * CKD Stage 3 (CKD-EPI eGFR ≥ 30 and < 60 mL/min/1.73 m2) and ONE or more of the following additional risk factors OR
   * CKD Stage 2 (CKD-EPI eGFR ≥ 60 and < 90 mL/min/1.73 m2) and ONE or more of the following additional risk factors:

     * Age ≥ 75 years;
     * Combined valve & coronary artery surgery;
     * Left ventricular ejection fraction (LVEF) ≤ 35% by invasive or noninvasive techniques;
     * Urinary (TIMP-2 x IGFBP7) > 0.3
     * Diabetes mellitus
     * Hypertension
     * Hyperlipidemia
4. Sexually active women of child-bearing potential (WCBP) must be using a medically acceptable method of birth control throughout the study and for at least 1 day following the end of study and have a negative urine pregnancy test at the Screening visit. A WCBP is defined as a female who is biologically capable of becoming pregnant. A medically acceptable method of birth control includes intrauterine devices in place for at least 3 months, surgical sterilization, or the implant. In patients who are not sexually active, abstinence is an acceptable form of birth control and urine will be tested per protocol. Women who are of nonchild-bearing potential, i.e., post-menopause, must have this condition captured in their medical history. Pregnant women and nursing mothers are excluded from this study.
5. Patient or Legally Authorized Representative (LAR) is available and willing to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.

Exclusion Criteria:

1. The presence of AKI (KDIGO criteria) at the time of randomization
2. Off-pump cardiac surgery
3. Surgery to be performed under conditions of circulatory arrest or hypothermia with rectal temperature < 28°C (82.4° F)
4. Severe chronic kidney disease: CKD-eGFR < 30 mL/min/1.73 m2) OR requiring dialysis
5. Imminent or recent surgery for aortic dissection
6. Surgery to correct a major congenital heart defect (e.g., Tetralogy of Fallot, transposition of the great vessels, single ventricle, or Ebstein's anomaly. Bicuspid aortic valve is not considered a congenital heart defect)
7. Known history of active cancer which may interfere with interpretation of the results of this study
8. Known or suspected sepsis at time of screening
9. Pregnancy or lactation
10. Known hypersensitivity to the study drug or any of its excipients
11. Treatment with an investigational drug or participation in an interventional trial within 30 days prior to the first dose of study drug and throughout the study
12. Any disease processes or confounding variables that would inappropriately alter the outcome of the study in the opinion of the investigator
13. Inability to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the percentage of subjects with AKI within 7 days following on-pump cardiac surgery defined by the KDIGO (Kidney Disease: Improving Global Outcomes) criteria | 7 days
  1. Increase in baseline (pre-surgery) serum creatinine (SCr) by ≥26.5 μmol/L (≥0.3 mg/dL) within 7 days; OR
  2. Increase in baseline SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the first 7 days following surgery; OR
  3. Urine output < 0.5 mL/kg/h for >6 hours.

SECONDARY OUTCOMES:
Maximum severity of AKI per patient between treatment groups | 7 days
  1. Stage 1: SCr 1.5 - 1.9 times baseline OR ≥26.5 μmol/L (≥0.3 mg/dL) increase OR urine output <0.5 mL/kg/hr for 6-12 hours
  2. Stage 2: SCr 2.0 - 2.9 times baseline OR urine output <0.5 mL/kg/h for ≥ 12 hours
  3. Stage 3: SCr ≥3.0 times baseline OR increase in SCr of ≥26.5 μmol/L (≥0.3 mg/dL) to ≥353.6 μmol/L (≥4.0 mg/dL) OR initiation of renal replacement therapy (RRT) OR urine output <0.3 mL/kg/h for ≥24 hours OR anuria for ≥12 hours.
Time to mild, moderate, and severe AKI per patient between treatment groups | 7 days
Need for RRT within the first 7 days following surgery | 7 days
Need for RRT at any time during the 28-day study | 28 days
Duration of AKI at 28 days (EOS) | 28 days
  Duration of AKI is defined as the number of days from start of AKI per KDIGO criteria to onset of resolution
Kidney function (SCr, eGFR) at 28 days (EOS) | 28 days
28-day all-cause mortality | 28 days
Composite of death, need for RRT, and/or persistent impaired renal function from baseline (MAKE [major adverse kidney event] criteria) at Day 28 (EOS) | 28 days
ICU length of stay (in days) | 28 days
Hospitalization length of stay (in days) | 28 days
Incidence of new-onset lung or liver disorders following surgery | 28 days
Change in baseline serum cystatin C, serum NGAL, serum IP-10, serum IL-1beta, serum IL-6, and serum IL-18 biomarker levels | 28 days
Changes in urinary TIMP-2 and IGFBP7 biomarker and serum NGAL, AGT, and IL-18 biomarker levels | 7 days
  Biomarkers will be measured at baseline and days 1, 3, 5, and 7
Development of serum anti-drug antibodies levels throughout the study | 28 days
  Anti-drug antibodies will be measured at baseline (Day 1 prior to the first dose of study medication) and at days 1, 2, 3, 4, 5 and day 28 (EOS)

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (4):
  - Cumming School of Medicine & Libin Cardiovascular Centre, University of Calgary, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
- Turkey (Türkiye) (5):
  - Gazi University, Yenimahalle, Ankara
  - Kosuyolu High Specialization Training and Research Hospital, Kartal, Istanbul
  - Erciyes University, Faculty of Medicine - Semiha Kibar Organ Transplant & Dialysis Hospital, Melikgazi, Kayseri
  - Kocaeli University, Faculty of Medicine Practices and Research Hospital, İzmit, Kocaeli
  - Sütçü İmam University, Faculty of Medicine, Kahramanmaraş, Onikişubat